CLINICAL TRIAL: NCT00235209
Title: A Study to Evaluate the Clinical Effectiveness of a Collagen-ORC Antimicrobial Matrix in Venous Leg Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 400-04-002
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2006-10

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

INTERVENTIONS:
Device: Collagen ORC Antimicrobial Matrix (CAM)

SUMMARY:
This is a randomized (1:1), prospective, open label, multicenter, comparative study to be examine the effectiveness of Collagen-ORC Antimicrobial matrix, a new wound dressing, on venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Have evidence of venous insufficiency documented by venous duplex scanning or impedance plethysmography within the past 6 months. The study report must contain the actual terms "venous incompetence" or it must be repeated.
* Have a venous ulcer of >3 but <25 cm2 in area, by planimetry.
* Have a venous ulcer that has been open continuously for >1 but <18 months prior to treatment.
* Have been in the prescribed compression for at least 7 days immediately prior to randomization, but no more than 14 days (consecutive or non-consecutive).
* If female, the subject must: be postmenopausal without menses for at least 1 year, or have had a hysterectomy or tubal ligation or otherwise be incapable of pregnancy, or have a negative serum Human Chorionic Gonadotropin (HCG) and be willing to practice an approved form of birth control for the duration of the trial.
* Subject agrees to participate in the study, including all study related procedures and evaluations and documents this agreement by signing the IRB-approved informed consent.

Exclusion Criteria:

* Have the designated study wound below the malleolus or above the popliteal fossa.
* Have been treated with becaplermin (PDGF-BB) or any other topical recombinant therapy to the study wound within the 30 days prior to randomization.
* Have had the study wound treated, at any time, with a skin substitute or an autologous growth factor.
* Have had a surgical procedure to treat venous or arterial disease of the affected limb within the past 90 days.
* Have evidence of significant arterial insufficiency (i.e. an ankle brachial index of < 0.8). Subjects with an ABI >1.0 must have a toe brachial index (TBI) of > 0.6 or a supine transcutaneous oxygen measurement on the affected leg and distal to the wound of >30mmHg.
* Have clinical evidence of active infection at the wound site.
* Have evidence of active vasculitis, cellulitis or collagen vascular disease.
* Have participated in a clinical trial of an investigational agent within the last 30 days.
* Have significant acute or chronic diseases (i.e., cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological or infectious diseases) that are not adequately controlled by medical treatment as determined by the Investigator's judgment.
* Have diabetes mellitus with a hemoglobin A1c > 10%.
* Have an active skin disease, such as psoriasis, which could impair the ability to assess the study wound.
* Have an allergy to the components of the dressings used in this study.
* Require concomitant use of pentoxifylline or clopidogrel bisulfate during the study.
* Have undergone enzymatic debridement of the study wound at any time during the 7 days prior to the first application of study treatment.
* Have any requirement for the use of systemic steroids or immunosuppressive or cytotoxic compounds during the period of the study or received low-dose steroid therapy for more than 5 days within the past year.
* Expect to undergo hyperbaric oxygen therapy at any time during the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-11; Study Completion 2005-12

PRIMARY OUTCOMES:
Clinical effectiveness of CAM in VLU by comparing the reduction in wound area during a 12-week treatment period.

SECONDARY OUTCOMES:
Effect of the 2 dressing regimens on rate of wound closure, ease of use, pain and adverse events, impact of the dressing regimen

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, MD, Study Director — Ethicon, Inc.
Locations (3):
- United States (3):
  - Wound Care Center, Fort Lauderdale, Florida
  - Foot and Ankle Institute of South Florida, South Miami, Florida
  - Penn North Centers for Advanced Wound Care, Warren, Pennsylvania